CLINICAL TRIAL: NCT03971721
Title: A Feasibility Study to Determine the Effects of a Novel Mattress Support for Treatment of Positional Obstructive Sleep Apnea at Home
Brief Title: Hill-Rom WAVE for Positional Obstructive Sleep Apnea at Home
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding stopped
Sponsor: Ohio State University (Other)
Collaborators: Hill-Rom (Industry)
Responsible Party: Principal Investigator, Ulysses Magalang MD, Principal Investigator, Ohio State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019H0025
Record Dates: First submitted 2019-05-30; First posted 2019-06-03 (Actual); Results first posted 2021-03-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-02

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Positional therapy
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Wave Mattress Support (Experimental): The mattress support will be delivered at the subject's home by professional staff of the sponsor (Hill-Rom) in the presence of the research coordinator or investigator. The subject will sleep on mattress support for the duration of study participation.
  Interventions: Device: Wave 4.3

INTERVENTIONS:
Device: Wave 4.3 — The Wave 4.3 mattress support is an insert, placed underneath the user's existing mattress, that when inflated increases the longitudinal incline of the mattress support, increasing in inclination in the direction of the head of the bed. The resulting mattress contours are such that the mattress has a lateral inclination of approximately 15 degrees in the head section and 10 degrees in the torso section. In addition to the features allowing the user to activate and deactivate creation of this Graduated Lateral RotationTM orientation, this device has sensors and monitoring system allowing for remotely monitoring the status of the system, including confirming that the supports are achieving the prescribed support angles, and that the system is working as planned.

SUMMARY:
1. Determine the effects of a mattress support (Wave 4.3) that promotes the avoidance of supine airway position at home on the apnea-hypopnea index (AHI) in patients with positional obstructive sleep apnea (OSA).
2. Determine the effects of Wave 4.3 on subjective measures of sleepiness and daytime function in patients with positional OSA.
3. Determine the effects of Wave 4.3 on subjective measures of sleep quality in patients with positional OSA.

DETAILED DESCRIPTION:
This is a preliminary single-arm study. The study will last up to 4 weeks including the screening period. Subjects will sleep using the mattress support at home for two consecutive weeks.

Outcome measures will include: AHI derived from HSAT (primary outcome), oxygen desaturation index (ODI), Epworth Sleepiness Scale (ESS) score, Functional Outcomes of Sleep Questionnaire (FOSQ), Visual Analog Scale (VAS) and questionnaire assessments of sleep quality, and actigraphic sleep measures. Subjects will also keep a sleep diary every night for the duration of the study. Subjects will be asked about their bed partners' report on snoring and witnessed apneas.

ELIGIBILITY:
Inclusion Criteria:

* • 18-75 years of age

  * Willing and able to give informed consent
  * Able to speak and understand English
  * Previous sleep study prior to enrollment done based on previous clinical evaluation by the subject's treating physician in the course of usual clinical care:

    1. overall AHI 5-40 events/hr.
    2. at least 10% time spent in the supine and 10% time in the non-supine positions.
    3. APOC I and APOC II
    4. central respiratory events < 50% of the total number of apneas and hypopneas
  * Using at least a queen-sized mattress when sleeping at home
  * Patients who meet the above criteria who have been prescribed CPAP or dental device but are non-adherent to treatment will be enrolled in the study. CPAP non-adherence will be defined as average nightly use < 4hrs/night based on a download of the CPAP machine, or self- acknowledged discontinuation or non-regular of CPAP use.

Exclusion Criteria:

* • Incapable of giving informed consent

  * Under the age of 18
  * Active titration of medication
  * Pregnancy, lactation (will be screened with urine pregnancy test)
  * Self-reported Substance abuse (current)
  * Excessive alcohol consumption

    * Excessive alcohol use is defined as:
    * More than 3 glasses of wine a day
    * More than 3 beers a day
    * More than 60 mL of hard liquor a day
  * Use of home oxygen
  * Presence of severe daytime sleepiness defined as an Epworth sleepiness scale score > 16 or a prior history of falling asleep while driving
  * Presence of cardiac pacemaker or automatic implantable cardioverter-defibrillator (AICD).
  * Unstable medical problem such as uncontrolled hypertension.
  * Body Mass Index (BMI) >45 kg/m2
  * Any other clinically significant condition that, in the opinion of the investigators, might put the subject at risk of harm during the study or might adversely affect the interpretation of the study data.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulysses Magalang, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Early termination of study by the sponsor limited the number of participants recruited.
Groups:
- Wave Mattress Support: The mattress support will be delivered at the subject's home by professional staff of the sponsor (Hill-Rom) in the presence of the research coordinator or investigator. Subject will sleep on mattress support for the duration of study participation.
  Wave 4.3: The Wave 4.3 mattress support is an insert, placed underneath the user's existing mattress, that when inflated increases the longitudinal incline of the mattress support, increasing in inclination in the direction of the head of the bed. The resulting mattress contours are such that the mattress has a lateral inclination of approximately 15 degrees in the head section and 10 degrees in the torso section. In addition to the features allowing the user to activate and deactivate creation of this Graduated Lateral RotationTM orientation, this device has sensors and monitoring system allowing for remotely monitoring the status of the system, including confirming that the supports are achieving the prescribed support angles and that the system is working as planned.
Period: Overall Study
Arm/Group | Wave Mattress Support
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Wave Mattress Support: The mattress support will be delivered at the subject's home by professional staff of the sponsor (Hill-Rom) in the presence of the research coordinator or investigator. Subject will sleep on mattress support for the duration of study participation.
  Wave 4.3: The Wave 4.3 mattress support is an insert, placed underneath the user's existing mattress, that when inflated increases the longitudinal incline of the mattress support, increasing in inclination in the direction of the head of the bed. The resulting mattress contours are such that the mattress has a lateral inclination of approximately 15 degrees in the head section and 10 degrees in the torso section. In addition to the features allowing the user to activate and deactivate creation of this Graduated Lateral RotationTM orientation, this device has sensors and monitoring system allowing for remotely monitoring the status of the system, including confirming that the supports are achieving the prescribed support angles, and that the system is working as planned.
Arm/Group | Wave Mattress Support
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 39.7 [33 to 46]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 3
Enrolled Participants [Count of Participants; unit: Participants] | 3

OUTCOME MEASURES:

1. Primary Outcome: Apnea-Hypopnea Index Difference Between Two Nights
Description: Apnea-Hypopnea Index derived from Home Sleep Test. The apnea-hypopnea index (AHI) is the combined average number of apneas and hypopneas that occur per hour of sleep between two nights. AHI<5 is indicative of no sleep apnea, AHI 5-15 is indicative of mild sleep apnea, AHI 15-30 is indicative of moderate sleep apnea, AHI>30 is indicative of severe sleep apnea. The minimum AHI is 0, and there is no maximum. A higher score means a worse outcome. Subscales are not used to compute the value. The difference was calculated based on the value at night 1 minus the value at night 2 (converted to a positive value if the difference created a negative value). The mean value was calculated by adding the difference based on the total number of participants.
Time Frame: 2 nights
Measure: Mean (Standard Deviation); unit: events per hour
Arm/Group | Wave Mattress Support
Number analyzed (Participants) | 3
events per hour | 2.03 (4.20)

2. Secondary Outcome: Oxygen Desaturation Index Difference Between Two Nights
Description: Oxygen Desaturation Index calculated based on the average between two nights measured. Desaturation episodes are generally described as a decrease in the mean oxygen saturation of ≥4% (over the last 120 seconds) that lasts for at least 10 seconds. ODI values can range from 0 to greater than 30. A higher score means a worse outcome. Subscales are not used to compute the value. The difference was calculated based on the value at night 1 minus the value at night 2 (converted to a positive value if the difference created a negative value). The mean value was calculated by adding the difference based on the total number of participants.
Time Frame: 2 nights
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Wave Mattress Support
Number analyzed (Participants) | 3
units on a scale | 1.33 (4.25)

3. Secondary Outcome: Epworth Sleepiness Score
Description: A subjective measure of sleepiness on average based on the total score. The score ranges from a minimum of 0 to a maximum of 24. A higher score means a worse outcome. Subscales are not used to compute the value. The difference was calculated based on the value at visit 1 minus the value at visit 4 (converted to a positive value if the difference created a negative value). The mean value was calculated by adding the difference based on the total number of participants.
Time Frame: Completed at Visit 1 and Visit 4 (~5 minutes)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Wave Mattress Support
Number analyzed (Participants) | 3
units on a scale | 6.67 (3.21)

4. Secondary Outcome: Functional Outcomes of Sleep Questionnaire Score
Description: A subjective measure of sleepiness on daytime function with an average of the total score. The score ranges from a minimum of 0 to a maximum of 20. A higher score means a better outcome. Subscales are not used to compute the value. The difference was calculated based on the value at visit 2 minus the value at visit 4 (converted to a positive value if the difference created a negative value). The difference was calculated based on the value at visit 2 minus the value at visit 4 (converted to a positive value if the difference created a negative value). The mean value was calculated by adding the difference based on the total number of participants.
Time Frame: Completed at Visit 2 and Visit 4 (~5 minutes)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Wave Mattress Support
Number analyzed (Participants) | 3
score on a scale | 2.00 (1.41)

5. Secondary Outcome: Visual Analog Scale Score
Description: A subjective measure of sleepiness with the average of the total score. The score ranges from a minimum of 0 to a maximum of 100. A higher score means a better outcome. Subscales are not used to compute the value. The difference was calculated based on the value at visit 2 minus the value at visit 4 (converted to a positive value if the difference created a negative value). The mean value was calculated by adding the difference based on the total number of participants.
Time Frame: Completed at Visit 2 and Visit 4 (~5 minutes)
Measure: Mean (Standard Deviation); unit: percentage of sleep quality
Arm/Group | Wave Mattress Support
Number analyzed (Participants) | 3
percentage of sleep quality | 34 (0)

ADVERSE EVENTS:
Time Frame: 4 months
Description: The participants in the study did not experience any adverse events. The study was terminated early by the sponsor before completion.
Arm/Group | Wave Mattress Support
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-12): https://cdn.clinicaltrials.gov/large-docs/21/NCT03971721/Prot_SAP_001.pdf